CLINICAL TRIAL: NCT00749944
Title: An Experimental Medicine, Randomized, Double-Blind Study Assessing Neuropsychiatric Symptoms In Quitting Smokers Treated With Varenicline Tartrate Or Placebo
Brief Title: Assessing Neuropsychiatric Symptoms Including Depression, Anxiety, Irritability, and Suicidal Thoughts or Behavior in Subjects Quitting Smoking on Varenicline Tartrate or Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3051115
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Results first posted 2010-08-09 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Smoking Cessation
Keywords: nicotine withdrawal, smoking cessation, varenicline
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- varenicline (Experimental)
  Interventions: Drug: varenicline
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — 1 mg tablets twice daily by mouth (after one week of uptitration: 0.5mg once daily for three days, 0.5mg twice daily for four days)
  Other Names: Chantix, Champix
  Arms: varenicline
Drug: placebo — 1 mg tablets twice daily by mouth (after one week of uptitration: 0.5mg once daily for three days, 0.5mg twice daily for four days)
  Arms: placebo

SUMMARY:
Study objective is to compare neuropsychiatric adverse events in subjects treated with varenicline or placebo in a controlled setting where both groups are experiencing nicotine withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* smokers who smoke >10 cigarettes/day and who have at least a moderate level of addiction as measured by the Fagerstrom Test for Nicotine Dependence (score >5)

Exclusion Criteria:

* Any neuropsychiatric disease including depression, history of suicidal thoughts or behavior, bipolar disorder.
* Any unstable medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- [Derived] Garza D, Murphy M, Tseng LJ, Riordan HJ, Chatterjee A. A double-blind randomized placebo-controlled pilot study of neuropsychiatric adverse events in abstinent smokers treated with varenicline or placebo. Biol Psychiatry. 2011 Jun 1;69(11):1075-82. doi: 10.1016/j.biopsych.2010.12.005. Epub 2011 Feb 3. PMID 21295286
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051115&StudyName=Assessing%20Neuropsychiatric%20Symptoms%20Including%20Depression%2C%20Anxiety%2C%20Irritability%2C%20and%20Suicidal%20Thoughts%20or%20Behavior%20in%20Subjects%20Quitting%20Sm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 857 participants were screened; 110 participants met the criteria for inclusion into the study and were assigned to study treatment
Groups:
- Varenicline: Varenicline 0.5 milligrams (mg) administered once daily (QD) for the first 3 days followed by 0.5 mg varenicline twice daily (BID) for the next 4 days, then 1 mg varenicline BID for the remaining 11 weeks (starting on Day 8, the first day of Week 2)
- Placebo: Placebo administered QD for the first 3 days followed by placebo administered BID for the remaining 11 weeks and 4 days (starting on Day 4)
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 55 | 55
Completed | 50 | 54
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Customized [Number; unit: Participants]
  Between 18 and 44 years | 47 | 47 | 94
  Between 45 and 64 years | 7 | 8 | 15
  >= 65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 37
  Male | 33 | 40 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Profile of Mood States (POMS): Total Mood Disturbance (TMD)
Description: POMS TMD were responses to 65 items in 6 subscales (Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor, Fatigue, and Confusion), on 'How you feel right now?' (scale:0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely). All items were rated in the same direction except for Relaxed and Efficient in the Tension-Anxiety and Confusion subscales. TMD was the sum of the scores of all 6 subscales but weighting Vigor negatively. Summary results (TMD scores) were presented as transformed T-scores ranging from 30 (less disturbance) to 80 (more disturbance).
Time Frame: Baseline A (Week 0) to Week 2 (Period AB), Week 4 (Period AC), Week 12 or relapse (Period AD), and Week 12 (Period AE). Baseline B (Week 2) to Week 4 (Period BC), Week 12 or relapse (Period BD), and Week 12 (Period BE).
Population: Full analysis set (FAS): All randomized subjects with at least 1 dose of study drug and at least 1 post-baseline neuropsychiatric evaluation or Minnesota Nicotine Withdrawal Scale (MNWS) obtained; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=55, 55) | 0.06 (0.39) | -0.66 (0.36)
  Period AC (n=55, 55) | 0.30 (0.35) | -0.17 (0.36)
  Period AD (n=55, 55) | 0.95 (0.43) | 0.03 (0.41)
  Period AE (n=55, 55) | 0.72 (0.36) | 0.22 (0.37)
  Period BC (n=53, 54) | 0.48 (0.35) | 0.91 (0.31)
  Period BD (n=53, 54) | 1.07 (0.47) | 1.04 (0.39)
  Period BE (n=54, 54) | 0.59 (0.37) | 0.96 (0.36)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.72, 95% CI 2-sided [-0.33 to 1.77]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.46, 95% CI 2-sided [-0.50 to 1.43]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.92, 95% CI 2-sided [-0.27 to 2.11]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.50, 95% CI 2-sided [-0.52 to 1.53]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.43, 95% CI 2-sided [-1.35 to 0.50] — Mixed Models Analysis
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.03, 95% CI 2-sided [-1.18 to 1.24]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.37, 95% CI 2-sided [-1.37 to 0.63] — Mixed Models Analysis

2. Primary Outcome: Change From Baseline in the Profile of Mood States (POMS): Tension-Anxiety Subscale
Description: POMS Tension-Anxiety subscale data were responses to 9 items regarding 'How you feel right now?' on a scale of 0=not at all, 1=a little, 2=moderately, 3=quite a bit, and 4=extremely. All items were rated in the same direction except for Relaxed. Summary results (subscale scores) were presented as transformed T-scores ranging from 30 (less disturbance) to 80 (more disturbance).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=55, 55) | 0.30 (0.30) | -0.31 (0.25)
  Period AC (n=55, 55) | 0.15 (0.25) | -0.26 (0.21)
  Period AD (n=55, 55) | 0.31 (0.24) | -0.18 (0.27)
  Period AE (n=55, 55) | 0.01 (0.24) | -0.43 (0.20)
  Period BC (n=53, 54) | -0.01 (0.24) | -0.10 (0.25)
  Period BD (n=53, 54) | 0.06 (0.23) | -0.16 (0.29)
  Period BE (n=54, 54) | -0.35 (0.19) | -0.58 (0.21)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.62, 95% CI 2-sided [-0.15 to 1.39]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.41, 95% CI 2-sided [-0.24 to 1.07]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.48, 95% CI 2-sided [-0.26 to 1.22]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.44, 95% CI 2-sided [-0.18 to 1.06]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.10, 95% CI 2-sided [-0.58 to 0.78]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.22, 95% CI 2-sided [-0.48 to 0.92]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.23, 95% CI 2-sided [-0.26 to 0.72]

3. Primary Outcome: Change From Baseline in the Profile of Mood States (POMS): Depression-Dejection Subscale
Description: POMS Depression-Dejection subscale data responses to 15 items regarding 'How you feel right now?' on a scale of 0=not at all, 1=a little, 2=moderately, 3=quite a bit, and 4=extremely. Summary results (subscale scores) were presented as transformed T-scores ranging from 30 (less disturbance) to 80 (more disturbance).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=55, 55) | 0.38 (0.25) | -0.24 (0.18)
  Period AC (n=55, 55) | 0.50 (0.24) | -0.24 (0.13)
  Period AD (n=55, 55) | 0.56 (0.27) | -0.10 (0.16)
  Period AE (n=55, 55) | 0.44 (0.24) | 0.00 (0.19)
  Period BC (n=53, 54) | 0.51 (0.27) | 0.03 (0.13)
  Period BD (n=53, 54) | 0.49 (0.32) | 0.10 (0.14)
  Period BE (n=54, 54) | 0.32 (0.23) | 0.23 (0.20)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.62, 95% CI 2-sided [-0.00 to 1.24]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.73, 95% CI 2-sided [0.18 to 1.29]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.66, 95% CI 2-sided [0.02 to 1.30]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.43, 95% CI 2-sided [-0.19 to 1.05]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.48, 95% CI 2-sided [-0.09 to 1.05]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.39, 95% CI 2-sided [-0.28 to 1.06]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.09, 95% CI 2-sided [-0.47 to 0.65]

4. Primary Outcome: Change From Baseline in the Profile of Mood States (POMS): Anger-Hostility Subscale
Description: POMS Anger-Hostility subscale data were responses to 12 items regarding 'How you feel right now?' on a scale of 0=not at all, 1=a little, 2=moderately, 3=quite a bit, and 4=extremely. Summary results (subscale scores) were presented as transformed T-scores ranging from 30 (less disturbance) to 80 (more disturbance).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=55, 55) | 0.16 (0.36) | -0.69 (0.25)
  Period AC (n=55, 55) | -0.04 (0.31) | -0.89 (0.16)
  Period AD (n=55, 55) | 0.24 (0.36) | -1.00 (0.22)
  Period AE (n=55, 55) | 0.15 (0.30) | -0.68 (0.15)
  Period BC (n=53, 54) | -0.00 (0.29) | -0.52 (0.15)
  Period BD (n=53, 54) | 0.22 (0.41) | -0.65 (0.19)
  Period BE (n=54, 54) | -0.05 (0.25) | -0.43 (0.18)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.85, 95% CI 2-sided [-0.02 to 1.72] — Mixed Models Analysis included baseline, treatment (t; fixed), subject (random), day (d; fixed), and interaction for t-by-d
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.85, 95% CI 2-sided [0.16 to 1.54] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 1.24, 95% CI 2-sided [0.39 to 2.08] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.83, 95% CI 2-sided [0.14 to 1.52] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.52, 95% CI 2-sided [-0.06 to 1.09] — Mixed Models Analysis included baseline, t (fixed), subject (random), time (fixed), d (fixed), and interactions for t-by-time, t-by-d, time-by-d and t-by-time-by-d
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.88, 95% CI 2-sided [0.05 to 1.70] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.38, 95% CI 2-sided [-0.12 to 0.88] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d

5. Primary Outcome: Change From Baseline in the Profile of Mood States (POMS): Vigor Subscale
Description: POMS Vigor subscale data were responses to 8 items regarding 'How you feel right now?' on a scale of 0=not at all, 1=a little, 2=moderately, 3=quite a bit, and 4=extremely. Summary results (subscale scores) were presented as transformed T-scores ranging from 30 (less disturbance) to 80 (more disturbance).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=55, 55) | 0.16 (0.86) | 0.98 (0.75)
  Period AC (n=55, 55) | -1.34 (0.87) | -1.15 (0.75)
  Period AD (n=55, 55) | -3.30 (1.18) | -1.14 (0.97)
  Period AE (n=55, 55) | -2.80 (1.00) | -1.82 (0.91)
  Period BC (n=53, 54) | -1.49 (0.81) | -3.44 (0.83)
  Period BD (n=53, 54) | -3.22 (1.25) | -3.22 (1.11)
  Period BE (n=54, 54) | -2.28 (1.02) | -3.37 (1.04)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.82, 95% CI 2-sided [-3.07 to 1.43] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.19, 95% CI 2-sided [-2.47 to 2.08] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -2.15, 95% CI 2-sided [-5.19 to 0.89] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.98, 95% CI 2-sided [-3.67 to 1.70] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 1.95, 95% CI 2-sided [-0.36 to 4.26] — [estimate comment as in outcome 4, analysis 5]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.01, 95% CI 2-sided [-3.32 to 3.30] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 1.09, 95% CI 2-sided [-1.80 to 3.97] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d

6. Primary Outcome: Change From Baseline in the Profile of Mood States (POMS): Fatigue Subscale
Description: POMS Fatigue subscale data were responses to 7 items regarding 'How you feel right now?' on a scale of 0=not at all, 1=a little, 2=moderately, 3=quite a bit, and 4=extremely. All items were rated in the same direction. Summary results (subscale scores) were presented as transformed T-scores ranging from 30 (less disturbance) to 80 (more disturbance).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=55, 55) | -0.14 (0.29) | -0.65 (0.29)
  Period AC (n=55, 55) | -0.29 (0.28) | -0.83 (0.24)
  Period AD (n=55, 55) | -0.58 (0.26) | -0.76 (0.27)
  Period AE (n=55, 55) | -0.32 (0.27) | -0.59 (0.24)
  Period BC (n=53, 54) | 0.37 (0.32) | -0.22 (0.23)
  Period BD (n=53, 54) | -0.20 (0.29) | -0.13 (0.30)
  Period BE (n=54, 54) | -0.16 (0.29) | -0.26 (0.25)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.52, 95% CI 2-sided [-0.29 to 1.32] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.54, 95% CI 2-sided [-0.17 to 1.25] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.18, 95% CI 2-sided [-0.55 to 0.92] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.26, 95% CI 2-sided [-0.46 to 0.99] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.59, 95% CI 2-sided [-0.19 to 1.37] — [estimate comment as in outcome 4, analysis 5]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.08, 95% CI 2-sided [-0.91 to 0.76] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.10, 95% CI 2-sided [-0.65 to 0.85] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d

7. Primary Outcome: Change From Baseline in the Profile of Mood States (POMS): Confusion Subscale
Description: POMS Confusion subscale data were responses to 7 items regarding 'How you feel right now?' on a scale of 0=not at all, 1=a little, 2=moderately, 3=quite a bit, and 4=extremely. All items were rated in the same direction except for Efficient. Summary results (subscale scores) were presented as transformed T-scores ranging from 30 (less disturbance) to 80 (more disturbance).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=55, 55) | 0.14 (0.19) | -0.09 (0.12)
  Period AC (n=55, 55) | 0.03 (0.17) | -0.18 (0.10)
  Period AD (n=55, 55) | 0.10 (0.18) | -0.11 (0.13)
  Period AE (n=55, 55) | -0.01 (0.15) | -0.03 (0.13)
  Period BC (n=53, 54) | 0.02 (0.22) | -0.07 (0.11)
  Period BD (n=53, 54) | 0.07 (0.22) | -0.02 (0.15)
  Period BE (n=54, 54) | -0.14 (0.18) | -0.02 (0.16)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.23, 95% CI 2-sided [-0.20 to 0.65] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.21, 95% CI 2-sided [-0.17 to 0.58] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.21, 95% CI 2-sided [-0.23 to 0.65] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.02, 95% CI 2-sided [-0.37 to 0.41] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.09, 95% CI 2-sided [-0.41 to 0.59] — [estimate comment as in outcome 4, analysis 5]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.10, 95% CI 2-sided [-0.44 to 0.63] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.12, 95% CI 2-sided [-0.58 to 0.34] — Mixed Models Analysis included baseline, t (fixed), subject (random), d (fixed), and interaction for t-by-d

8. Primary Outcome: Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS): Total Score
Description: The MADRS measures the overall severity of depressive symptoms and is a 10-item checklist. Each item was rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | 1.05 (0.37) | 0.83 (0.25)
  Period AC (n=54, 54) | 2.28 (0.35) | 1.84 (0.30)
  Period AD (n=54, 54) | 1.19 (0.29) | 1.41 (0.37)
  Period AE (n=55, 54) | 1.52 (0.21) | 1.50 (0.28)
  Period BC (n=53, 54) | 2.27 (0.50) | 1.69 (0.48)
  Period BD (n=53, 54) | -0.10 (0.35) | 0.33 (0.53)
  Period BE (n=53, 54) | 0.40 (0.24) | 0.49 (0.30)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.22, 95% CI 2-sided [-0.66 to 1.10] — Mixed Models Analysis included baseline, treatment (fixed effect), subject (random effect), week (fixed effect), and interaction of treatment-by-week
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.44, 95% CI 2-sided [-0.46 to 1.35] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.22, 95% CI 2-sided [-1.16 to 0.71] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.03, 95% CI 2-sided [-0.68 to 0.73] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.58, 95% CI 2-sided [-0.79 to 1.96] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.43, 95% CI 2-sided [-1.69 to 0.82] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.09, 95% CI 2-sided [-0.86 to 0.68] — [estimate comment as in outcome 8, analysis 1]

9. Primary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A): Total Score
Description: HAM-A measures treatment-related changes in generalized anxiety symptoms and is a 14-item questionnaire. Each item was scored from 0 (not present) to 4 (very severe) and a lower score indicated less affected. Total scores ranged from 0 (not affected) to 56 (very severely affected).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | 1.01 (0.32) | 0.75 (0.27)
  Period AC (n=54, 54) | 2.69 (0.37) | 2.16 (0.28)
  Period AD (n=54, 54) | 1.95 (0.41) | 1.86 (0.42)
  Period AE (n=55, 54) | 1.75 (0.28) | 1.61 (0.26)
  Period BC (n=53, 54) | 3.15 (0.56) | 2.65 (0.47)
  Period BD (n=53, 54) | 0.74 (0.47) | 0.77 (0.62)
  Period BE (n=53, 54) | 0.73 (0.30) | 0.81 (0.29)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.27, 95% CI 2-sided [-0.55 to 1.08] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.53, 95% CI 2-sided [-0.39 to 1.46] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.09, 95% CI 2-sided [-1.08 to 1.25] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.14, 95% CI 2-sided [-0.62 to 0.90] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.50, 95% CI 2-sided [-0.94 to 1.95] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.03, 95% CI 2-sided [-1.57 to 1.51] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.08, 95% CI 2-sided [-0.91 to 0.75] — [estimate comment as in outcome 8, analysis 1]

10. Primary Outcome: Change From Baseline in the Overt Aggression Scale (Modified) (OAS-m): Aggression Total Score
Description: The OAS-m contains 3 scales: Aggression (Questions [Q]1 to 4), Irritability (Q5 to 6), and Suicidality (Q7 to 7b). Aggression total score was calculated by summing the weighted scores in Q1 to 4. Scores for each question ranged from 0 (no events) to 5 (very severe events). Total scores ranged from 0 (no aggression) to any number with no upper limit depending on the frequency of agressive behaviour in a week.
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | 0.13 (0.27) | 0.48 (0.66)
  Period AC (n=54, 54) | 0.82 (0.37) | 0.72 (0.39)
  Period AD (n=54, 54) | 2.24 (1.75) | 0.75 (0.34)
  Period AE (n=55, 54) | 1.27 (0.70) | 0.77 (0.48)
  Period BC (n=53, 54) | 0.83 (0.63) | 0.22 (0.38)
  Period BD (n=53, 54) | 1.94 (2.27) | -0.15 (0.44)
  Period BE (n=53, 54) | 1.00 (0.88) | -0.13 (0.23)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.35, 95% CI 2-sided [-1.76 to 1.06] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.11, 95% CI 2-sided [-0.96 to 1.17] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 1.49, 95% CI 2-sided [-1.94 to 4.91] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.50, 95% CI 2-sided [-1.18 to 2.18] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.61, 95% CI 2-sided [-0.85 to 2.07] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 2.10, 95% CI 2-sided [-2.60 to 6.79] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 1.13, 95% CI 2-sided [-0.70 to 2.96] — [estimate comment as in outcome 8, analysis 1]

11. Primary Outcome: Change From Baseline in the Overt Aggression Scale (Modified) (OAS-m): Irritability Total Score
Description: The OAS-m contains 3 scales: Aggression (Questions [Q]1 to 4), Irritability (Q5 to 6), and Suicidality (Q7 to 7b). Irritability total score was calculated by summing the items in Q5 to 6. Scores for each question ranged from 0 (not at all) to 5 (extreme). Total scores ranged from 0 (no irritability) to 10 (extreme irritability).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | 0.01 (0.10) | 0.01 (0.09)
  Period AC (n=54, 54) | 0.43 (0.10) | 0.41 (0.09)
  Period AD (n=54, 54) | 0.46 (0.17) | 0.35 (0.17)
  Period AE (n=55, 54) | 0.32 (0.10) | 0.24 (0.08)
  Period BC (n=53, 54) | 0.82 (0.16) | 0.78 (0.16)
  Period BD (n=53, 54) | 0.53 (0.19) | 0.35 (0.24)
  Period BE (n=53, 54) | 0.38 (0.11) | 0.25 (0.08)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.00, 95% CI 2-sided [-0.26 to 0.27] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.02, 95% CI 2-sided [-0.25 to 0.29] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.10, 95% CI 2-sided [-0.37 to 0.58] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.08, 95% CI 2-sided [-0.17 to 0.34] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.04, 95% CI 2-sided [-0.40 to 0.48] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.17, 95% CI 2-sided [-0.44 to 0.78] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.13, 95% CI 2-sided [-0.14 to 0.40] — [estimate comment as in outcome 8, analysis 1]

12. Primary Outcome: Change From Baseline in the Overt Aggression Scale (Modified) (OAS-m): Suicidality Total Score
Description: The OAS-m contains 3 scales: Aggression (Questions [Q]1 to 4), Irritability (Q5 to 6), and Suicidality (Q7 to 7b). Suicidality total score was calculated by summing the items Q7 to 7b. Scores for Q7 ranged from 0 (none) to 6 (very extreme) and scores for Q7a to 7b ranged from 0 (none) to 5 (extreme). Total scores ranged from 0 (no suicidal tendency) to 16 (extreme/very extreme suicidal tendency).
Time Frame: as for outcome 1
Population: No change from baseline analysis was performed on the OAS-m Suicidality total score as the majority of observations were recorded as 0.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Change From Baseline in the Social Dysfunction and Aggression Scale (SDAS): Total Score
Description: The SDAS contains 11 items with 5 possible responses: 0=not present, 1=doubtful or very mild, 2=mild to moderate, 3=severe, and 4=extremely severe. The SDAS was collected 3 times a day during the inpatient abstinence period (BC). Total scores ranged from 0 (not present) to 44 (extremely severe).
Time Frame: Baseline B (Week 2) to Week 4 (Period BC)
Population: No change from baseline analysis was performed on the SDAS total score as the majority of observations were recorded as 0.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Change From Baseline in the Barratt Impulsiveness Scale - Version 11 (BIS-11): Total Score
Description: The BIS-11 is a 30-item self-report questionnaire designed to assess general impulsiveness taking into account the multifactorial nature of the construct. Possible responses to each item were: 1=rarely/never, 2=occasionally, 3=often, and 4=almost always/always. Scores of Items 1, 7, 8, 9, 10, 12, 13, 15, 20, 29 and 30 were reversed when calculating the total score. Total score ranged from 30 (less impulsive) to 120 (more impulsive).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | 0.34 (0.56) | -0.07 (0.50)
  Period AC (n=54, 54) | 0.45 (0.62) | 0.37 (0.53)
  Period AD (n=54, 54) | 1.34 (0.74) | 1.28 (1.03)
  Period AE (n=55, 54) | 1.19 (0.69) | 0.90 (0.64)
  Period BC (n=53, 54) | 0.04 (0.49) | 0.97 (0.43)
  Period BD (n=53, 54) | 1.07 (0.49) | 1.81 (0.92)
  Period BE (n=53, 54) | 0.85 (0.52) | 1.28 (0.44)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.41, 95% CI 2-sided [-1.09 to 1.90] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.08, 95% CI 2-sided [-1.54 to 1.71] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.06, 95% CI 2-sided [-2.47 to 2.60] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.29, 95% CI 2-sided [-1.57 to 2.15] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.94, 95% CI 2-sided [-2.23 to 0.36] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.74, 95% CI 2-sided [-2.81 to 1.33] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.43, 95% CI 2-sided [-1.78 to 0.92] — [estimate comment as in outcome 8, analysis 1]

15. Secondary Outcome: Change From Baseline in the Minnesota Nicotine Withdrawal Scale (MNWS): Total Score
Description: The MNWS total score contains 9 items (urge to smoke; depressed mood; irritability, frustration, or anger; anxiety; difficulty concentrating; restlessness; increased appetite; difficulty going to sleep; difficulty staying asleep). Each item was rated from 0 to 4 where 0=not at all, 1=slight, 2=moderate, 3=quite a bit, and 4=extreme. Total scores were the average score for all 9 items and ranged from 0 (no withdrawal symptoms) to 4 (extreme withdrawal symptoms).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | 0.13 (0.04) | 0.05 (0.04)
  Period AC (n=54, 54) | 0.10 (0.03) | 0.11 (0.03)
  Period AD (n=54, 54) | 0.07 (0.03) | 0.05 (0.03)
  Period AE (n=55, 54) | -0.01 (0.02) | 0.04 (0.03)
  Period BC (n=53, 54) | -0.04 (0.04) | 0.10 (0.06)
  Period BD (n=53, 54) | -0.08 (0.03) | 0.02 (0.04)
  Period BE (n=53, 54) | -0.15 (0.01) | -0.05 (0.03)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.08, 95% CI 2-sided [-0.04 to 0.19] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.01, 95% CI 2-sided [-0.11 to 0.08] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.02, 95% CI 2-sided [-0.06 to 0.09] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.05, 95% CI 2-sided [-0.11 to 0.02] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.14, 95% CI 2-sided [-0.27 to -0.01] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.10, 95% CI 2-sided [-0.21 to 0.01] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.10, 95% CI 2-sided [-0.17 to -0.03] — [estimate comment as in outcome 8, analysis 1]

16. Secondary Outcome: Change From Baseline in the Minnesota Nicotine Withdrawal Scale (MNWS): Negative Affect Domain Subscale
Description: The MNWS negative affect domain subscale contains 4 items (depressed mood; irritability, frustration, or anger; anxiety; difficulty concentrating). Each item was rated from 0 to 4 where 0=not at all, 1=slight, 2=moderate, 3=quite a bit, and 4=extreme. Scores were the average from all 4 items and ranged from 0 (no negative affect) to 4 (extreme negative affect).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | 0.06 (0.03) | 0.01 (0.02)
  Period AC (n=54, 54) | 0.10 (0.03) | 0.09 (0.03)
  Period AD (n=54, 54) | 0.07 (0.03) | 0.03 (0.03)
  Period AE (n=55, 54) | 0.05 (0.02) | 0.07 (0.03)
  Period BC (n=53, 54) | 0.07 (0.05) | 0.15 (0.05)
  Period BD (n=53, 54) | -0.01 (0.03) | 0.02 (0.05)
  Period BE (n=53, 54) | -0.02 (0.02) | 0.03 (0.03)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.05, 95% CI 2-sided [-0.03 to 0.12] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.00, 95% CI 2-sided [-0.08 to 0.09] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.03, 95% CI 2-sided [-0.04 to 0.11] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.01, 95% CI 2-sided [-0.08 to 0.05] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.08, 95% CI 2-sided [-0.22 to 0.06] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.03, 95% CI 2-sided [-0.14 to 0.09] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.05, 95% CI 2-sided [-0.11 to 0.02] — [estimate comment as in outcome 8, analysis 1]

17. Secondary Outcome: Change From Baseline in the Minnesota Nicotine Withdrawal Scale (MNWS): Insomnia Domain Subscale
Description: The MNWS insomnia domain subscale contains 2 items (difficulty going to sleep; difficulty staying asleep). Each item was rated from 0 to 4 where 0=not at all, 1=slight, 2=moderate, 3=quite a bit, and 4=extreme. Scores were the average of the 2 items and ranged from 0 (no insomnia) to 4 (extreme insomnia).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | 0.07 (0.04) | 0.12 (0.06)
  Period AC (n=54, 54) | 0.15 (0.04) | 0.17 (0.05)
  Period AD (n=54, 54) | 0.04 (0.03) | 0.10 (0.04)
  Period AE (n=55, 54) | 0.06 (0.02) | 0.13 (0.06)
  Period BC (n=53, 54) | 0.14 (0.07) | 0.09 (0.08)
  Period BD (n=53, 54) | -0.04 (0.05) | 0.01 (0.06)
  Period BE (n=53, 54) | -0.06 (0.02) | -0.01 (0.06)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.06, 95% CI 2-sided [-0.20 to 0.09] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.02, 95% CI 2-sided [-0.15 to 0.12] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.05, 95% CI 2-sided [-0.15 to 0.04] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.08, 95% CI 2-sided [-0.20 to 0.04] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.05, 95% CI 2-sided [-0.17 to 0.27] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.05, 95% CI 2-sided [-0.21 to 0.10] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.05, 95% CI 2-sided [-0.17 to 0.07] — [estimate comment as in outcome 8, analysis 1]

18. Secondary Outcome: Change From Baseline in the Minnesota Nicotine Withdrawal Scale (MNWS): Urge to Smoke Subscale
Description: The MNWS urge to smoke subscale contains 1 item (urge to smoke) rated from 0 to 4 where 0=not at all, 1=slight, 2=moderate, 3=quite a bit, and 4=extreme. Scores ranged from 0 (no urge to smoke) to 4 (extreme urge to smoke).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | -0.60 (0.10) | -0.29 (0.09)
  Period AC (n=54, 54) | -1.40 (0.09) | -0.97 (0.09)
  Period AD (n=54, 54) | -2.17 (0.12) | -2.03 (0.12)
  Period AE (n=55, 54) | -1.90 (0.09) | -1.55 (0.09)
  Period BC (n=53, 54) | -1.59 (0.12) | -1.14 (0.14)
  Period BD (n=53, 54) | -1.66 (0.14) | -1.58 (0.15)
  Period BE (n=53, 54) | -1.56 (0.10) | -1.29 (0.11)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline = -0.30, 95% CI 2-sided [-0.58 to -0.02] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline = -0.44, 95% CI 2-sided [-0.69 to -0.19] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline = -0.14, 95% CI 2-sided [-0.47 to 0.20] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline = -0.35, 95% CI 2-sided [-0.61 to -0.09] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline = -0.45, 95% CI 2-sided [-0.83 to -0.07] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline = -0.08, 95% CI 2-sided [-0.50 to 0.34] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline = -0.27, 95% CI 2-sided [-0.57 to 0.02] — [estimate comment as in outcome 8, analysis 1]

19. Secondary Outcome: Change From Baseline in the Minnesota Nicotine Withdrawal Scale (MNWS): Restlessness Subscale
Description: The MNWS restlessness subscale contains 1 item (restlessness) rated from 0 to 4 where 0=not at all, 1=slight, 2=moderate, 3=quite a bit, and 4=extreme. Scores ranged from 0 (no restlessness) to 4 (extreme restlessness).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | 0.06 (0.04) | 0.08 (0.04)
  Period AC (n=54, 54) | 0.10 (0.04) | 0.11 (0.04)
  Period AD (n=54, 54) | 0.09 (0.04) | 0.04 (0.03)
  Period AE (n=55, 54) | 0.03 (0.02) | 0.05 (0.03)
  Period BC (n=53, 54) | 0.07 (0.05) | 0.08 (0.05)
  Period BD (n=53, 54) | 0.03 (0.02) | -0.03 (0.01)
  Period BE (n=53, 54) | -0.04 (0.02) | -0.03 (0.03)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.02, 95% CI 2-sided [-0.12 to 0.08] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.02, 95% CI 2-sided [-0.12 to 0.08] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.05, 95% CI 2-sided [-0.04 to 0.14] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.01, 95% CI 2-sided [-0.07 to 0.04] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.01, 95% CI 2-sided [-0.15 to 0.13] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.06, 95% CI 2-sided [0.01 to 0.10] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.02, 95% CI 2-sided [-0.08 to 0.04] — [estimate comment as in outcome 8, analysis 1]

20. Secondary Outcome: Change From Baseline in the Minnesota Nicotine Withdrawal Scale (MNWS): Increased Appetite Subscale
Description: The MNWS increased appetite subscale contains 1 item (increased appetite) rated from 0 to 4 where 0=not at all, 1=slight, 2=moderate, 3=quite a bit, and 4=extreme. Scores ranged from 0 (no increased appetite) to 4 (extreme increased appetite).
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
scores on a scale
  Period AB (n=54, 54) | 0.14 (0.07) | 0.02 (0.05)
  Period AC (n=54, 54) | 0.10 (0.05) | 0.12 (0.06)
  Period AD (n=54, 54) | 0.11 (0.09) | 0.15 (0.09)
  Period AE (n=55, 54) | -0.00 (0.05) | 0.04 (0.06)
  Period BC (n=53, 54) | -0.03 (0.07) | 0.16 (0.08)
  Period BD (n=53, 54) | -0.01 (0.09) | 0.15 (0.10)
  Period BE (n=53, 54) | -0.10 (0.04) | -0.03 (0.06)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = 0.12, 95% CI 2-sided [-0.05 to 0.28] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.02, 95% CI 2-sided [-0.19 to 0.14] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.04, 95% CI 2-sided [-0.29 to 0.22] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.04, 95% CI 2-sided [-0.20 to 0.13] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.19, 95% CI 2-sided [-0.40 to 0.01] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.16, 95% CI 2-sided [-0.42 to 0.10] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo; Test type: Superiority or Other; Difference (change from baseline) = -0.07, 95% CI 2-sided [-0.22 to 008] — [estimate comment as in outcome 8, analysis 1]

21. Secondary Outcome: Number of Participants Exceeding Thresholds for the Profile of Mood States (POMS): Total Score
Description: POMS total mood disturbance (TMD) summary results were presented as transformed T-scores ranging from 30 (less disturbance) to 80 (more disturbance). Participants exceeding the threshold had an increase from baseline of 1 standard deviation of the TMD baseline T-score plus 1 or more.
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
participants
  Period AB (n=55, 55) | 14 | 11
  Period AC (n=55, 55) | 32 | 35
  Period AD (n=55, 55) | 37 | 38
  Period AE (n=55, 55) | 38 | 38
  Period BC (n=53, 54) | 27 | 33
  Period BD (n=53, 54) | 30 | 36
  Period BE (n=54, 54) | 32 | 38
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AB: Difference varenicline versus placebo. Subjects' worst scores observed in a given period were compared with the threshold criterion for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.6 to 3.3] — Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Period AC: Difference varenicline versus placebo. Subjects' worst scores observed in a given period were compared with the threshold criterion for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.7] — Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Period AD: Difference varenicline versus placebo. Subjects' worst scores observed in a given period were compared with the threshold criterion for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.4 to 2.1] — Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Period AE: Difference varenicline versus placebo. Subjects' worst scores observed in a given period were compared with the threshold criterion for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.4 to 2.2] — Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Period BC: Difference varenicline versus placebo. Subjects' worst scores observed in a given period were compared with the threshold criterion for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.3 to 1.4] — Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Period BD: Difference varenicline versus placebo. Subjects' worst scores observed in a given period were compared with the threshold criterion for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.3 to 1.4] — Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Period BE: Difference varenicline versus placebo. Subjects' worst scores observed in a given period were compared with the threshold criterion for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.3 to 1.4] — Cochran-Mantel-Haenszel

22. Secondary Outcome: Number of Participants Exceeding Thresholds for the Montgomery-Asberg Depression Rating Scale (MADRS): Total Score
Description: The MADRS measures the overall severity of depressive symptoms. Total score ranged from 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Participants exceeding the threshold had a MADRS total score of more than 14 out of 60. MADRS total scores exceeding 14 may represent clinically notable effective symptomatology.
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively. Statistical analyses were not performed for Period AB due to the small number of participants exceeding the threshold.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
participants
  Period AB (n=54, 54) | 2 | 0
  Period AC (n=54, 54) | 7 | 3
  Period AD (n=54, 54) | 8 | 3
  Period AE (n=55, 54) | 11 | 8
  Period BC (n=53, 54) | 5 | 3
  Period BD (n=53, 54) | 6 | 3
  Period BE (n=54, 54) | 9 | 8
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period AC: Difference varenicline versus placebo. Subjects' worst scores observed in a given period were compared with the threshold criterion for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 2.5, 95% CI 2-sided [0.6 to 10.4] — Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority or Other; Odds Ratio (OR) = 3.0, 95% CI 2-sided [0.7 to 11.8] — Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.5 to 3.9] — Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority or Other; Odds Ratio (OR) = 1.8, 95% CI 2-sided [0.4 to 7.8] — Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority or Other; Odds Ratio (OR) = 2.2, 95% CI 2-sided [0.5 to 9.2] — Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority or Other; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.4 to 3.2] — Cochran-Mantel-Haenszel

23. Secondary Outcome: Number of Participants Exceeding Thresholds for the Hamilton Anxiety Scale (HAM-A): Total Score
Description: HAM-A measures treatment-related changes in generalized anxiety symptoms. Total scores ranged from 0 (not affected) to 56 (very severely affected). Participants exceeding the threshold had a HAM-A total score of more than or equal to 14 out of 56. HAM-A total scores of more than or equal to 14 may reflect clinically noteworthy levels of anxiety.
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
participants
  Period AB (n=54, 54) | 0 | 2
  Period AC (n=54, 54) | 9 | 7
  Period AD (n=54, 54) | 12 | 7
  Period AE (n=55, 54) | 16 | 10
  Period BC (n=53, 54) | 9 | 6
  Period BD (n=53, 54) | 12 | 6
  Period BE (n=54, 54) | 16 | 9
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 2]; Test type: Superiority or Other; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.5 to 3.9] — Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority or Other; Odds Ratio (OR) = 1.9, 95% CI 2-sided [0.7 to 5.3] — Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; Odds Ratio (OR) = 1.8, 95% CI 2-sided [0.7 to 4.4] — Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority or Other; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.5 to 5.0] — Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority or Other; Odds Ratio (OR) = 2.3, 95% CI 2-sided [0.8 to 6.8] — Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority or Other; Odds Ratio (OR) = 2.1, 95% CI 2-sided [0.8 to 5.3] — Cochran-Mantel-Haenszel

24. Secondary Outcome: Number of Participants Exceeding Thresholds for the Overt Aggression Scale (Modified) (OAS-m): Agression Total Score
Description: The OAS-m contains 3 scales: Aggression, Irritability, and Suicidality. Aggression total score ranged from 0 (no aggression) to any number with no upper limit depending on the frequency of agressive behaviour in a week. Participants exceeding the threshold had an OAS-m Aggression total score of more than or equal to 3 out of any number with no upper limit depending on the frequency of agressive behaviour in a week. OAS-m Aggression total scores of more than or equal to 3 reflect clinically important aggression.
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
participants
  Period AB (n=54, 54) | 9 | 6
  Period AC (n=54, 54) | 20 | 21
  Period AD (n=54, 54) | 21 | 23
  Period AE (n=55, 54) | 28 | 31
  Period BC (n=53, 54) | 15 | 19
  Period BD (n=53, 54) | 18 | 21
  Period BE (n=54, 54) | 27 | 30
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.5 to 4.9] — Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 2]; Test type: Superiority or Other; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.4 to 2.0] — Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority or Other; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.4 to 1.8] — Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.6] — Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority or Other; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.3 to 1.6] — Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority or Other; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.8] — Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority or Other; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.7] — Cochran-Mantel-Haenszel

25. Secondary Outcome: Number of Participants Exceeding Thresholds for the Overt Aggression Scale (Modified) (OAS-m): Irritability Total Score
Description: The OAS-m contains 3 scales: Aggression, Irritability, and Suicidality. Irritability total score ranged from 0 (no irritability) to 10 (extreme irritability). Participants exceeding the threshold had an OAS-m Irritability total score of more than or equal to 2 out of 10. OAS-m Irritability total scores of more than or equal to 2 reflect clinically important irritability.
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
participants
  Period AB (n=54, 54) | 10 | 11
  Period AC (n=54, 54) | 32 | 34
  Period AD (n=54, 54) | 36 | 36
  Period AE (n=55, 54) | 41 | 39
  Period BC (n=53, 54) | 31 | 31
  Period BD (n=53, 54) | 35 | 33
  Period BE (n=54, 54) | 40 | 38
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.3 to 2.3] — Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 2]; Test type: Superiority or Other; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.4 to 1.9] — Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority or Other; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.4 to 2.2] — Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.5 to 2.6] — Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority or Other; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.5 to 2.3] — Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority or Other; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.6 to 2.7] — Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority or Other; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.5 to 2.8] — Cochran-Mantel-Haenszel

26. Secondary Outcome: Number of Participants Exceeding Thresholds for the Overt Aggression Scale (Modified) (OAS-m): Suicidality Total Score
Description: The OAS-m contains 3 scales: Aggression, Irritability, and Suicidality. Suicidality total score ranged from 0 (no suicidal tendency) to 16 (extreme/very extreme suicidal tendency). No threshold criterion was determined for OAS-m Suicidality total score.
Time Frame: as for outcome 1
Population: The number of participants above the threshold for the OAS-m Suicidality total score was not analyzed as the majority of observations were recorded as 0.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Number of Participants Exceeding Thresholds for the Barratt Impulsiveness Scale - Version 11 (BIS-11): Total Score
Description: The BIS-11 is designed to assess general impulsiveness taking into account the multifactorial nature of the construct. Total score ranged from 30 (less impulsive) to 120 (more impulsive). Participants exceeding the threshold had a BIS-11 total score more than or equal to 70 out of 120. BIS-11 total scores of more than or equal to 70 could reflect clinically important and potentially pathological impulsivity.
Time Frame: as for outcome 1
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
participants
  Period AB (n=54, 54) | 1 | 0
  Period AC (n=54, 54) | 1 | 2
  Period AD (n=54, 54) | 1 | 2
  Period AE (n=55, 54) | 5 | 5
  Period BC (n=53, 54) | 1 | 2
  Period BD (n=53, 54) | 1 | 2
  Period BE (n=54, 54) | 5 | 5
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.0 to 5.6] — Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 3]; Test type: Superiority or Other; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.0 to 5.6] — Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.3 to 3.6] — Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 5]; Test type: Superiority or Other; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.0 to 5.7] — Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 6]; Test type: Superiority or Other; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.0 to 5.7] — Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Varenicline vs Placebo; [analysis description as in outcome 21, analysis 7]; Test type: Superiority or Other; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.3 to 3.7] — Cochran-Mantel-Haenszel

28. Secondary Outcome: Number of Participants Exceeding Thresholds for the Social Dysfunction and Aggression Scale (SDAS): Total Score
Description: SDAS total scores ranged from 0 (not present) to 44 (extremely severe). Participants exceeding the threshold had a SDAS total score of more than 6 out of 44.
Time Frame: Baseline B (Week 2) to Week 4 (Period BC)
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
participants | 2 | 1
Statistical Analysis 1: Comparison: Varenicline vs Placebo; There was no hypothesis testing or power calculation in this study. Period BC: Difference varenicline versus placebo. Subjects' worst scores observed in a given period were compared with the threshold criterion for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 2.1, 95% CI 2-sided [0.2 to 23.6] — Cochran-Mantel-Haenszel

29. Secondary Outcome: Number of Participants With Carbon Monoxide Confirmed Daily Smoking Cessation
Description: Participants who reported no smoking and no use of other nicotine-containing products since the last study visit (on the Nicotine Use Inventory, which was used to collect the information of cigarette or other nicotine use during the study) and who did not have carbon monoxide of more than 10 parts per million at any time from Week 9 to Week 12
Time Frame: Week 9 to Week 12
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
participants | 16 | 10

30. Secondary Outcome: Number of Participants With 7-day Point Prevalence of Abstinence (Smoking Cessation)
Description: Participants who reported no smoking and no use of other nicotine-containing products since the last study visit (during treatment) in the previous 7 days and who did not have carbon monoxide of more than 10 parts per million for that observation (if measured).
Time Frame: Week 5 to Week 13
Population: FAS; (n)=number of subjects with data for analysis for varenicline and placebo, respectively.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
participants
  Week 5 (n=55, 55) | 19 | 16
  Week 6 (n=55, 55) | 23 | 12
  Week 7 (n=55, 55) | 20 | 17
  Week 8 (n=55, 55) | 21 | 15
  Week 9 (n=55, 55) | 25 | 14
  Week 10 (n=55, 55) | 17 | 17
  Week 11 (n=55, 55) | 20 | 18
  Week 12 (n=55, 55) | 19 | 15
  Week 13 (n=55, 55) | 23 | 15

31. Secondary Outcome: Change From Baseline in the Number of Cigarettes Smoked Per Day
Time Frame: Baseline (Week 0) to Week 2
Population: FAS; (n)=number of subjects with at least 1 dose of study drug and an observation for a given day.
Measure: Mean (Standard Deviation); unit: cigarettes smoked per day
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 55 | 55
cigarettes smoked per day
  Day 2 (n=55, 54) | -0.1 (3.6) | -0.2 (3.7)
  Day 3 (n=55, 54) | -0.6 (4.1) | 0.0 (3.9)
  Day 4 (n=55, 54) | -1.8 (5.0) | -0.3 (3.7)
  Day 5 (n=55, 54) | -1.0 (5.2) | -0.4 (4.0)
  Day 6 (n=54, 54) | -1.3 (5.9) | 0.1 (4.5)
  Day 7 (n=54, 54) | -1.8 (4.9) | -0.3 (5.0)
  Day 8 (n=54, 54) | -1.7 (5.0) | 0.4 (4.3)
  Day 9 (n=52, 54) | -1.0 (5.1) | 0.1 (4.2)
  Day 10 (n=52, 54) | -1.7 (5.7) | -0.4 (6.1)
  Day 11 (n=53, 54) | -1.8 (5.3) | -0.4 (6.3)
  Day 12 (n=53, 54) | -0.7 (6.6) | -0.2 (6.3)
  Day 13 (n=53, 54) | -1.4 (5.6) | -0.1 (6.1)
  Day 14 (n=36, 38) | -17.2 (8.6) | -15.7 (6.6)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 54/55 | 52/55
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=55) | Placebo (N=55)
Palpitations (Cardiac disorders) | 2 | 3
Ear pain (Ear and labyrinth disorders) | 4 | 2
Tinnitus (Ear and labyrinth disorders) | 3 | 2
Conjunctival irritation (Eye disorders) | 0 | 2
Eye irritation (Eye disorders) | 1 | 3
Vision blurred (Eye disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 10 | 5
Abdominal tenderness (Gastrointestinal disorders) | 2 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 2
Chapped lips (Gastrointestinal disorders) | 10 | 7
Constipation (Gastrointestinal disorders) | 8 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 5 | 1
Flatulence (Gastrointestinal disorders) | 3 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 18 | 16
Toothache (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 7 | 5
Asthenia (General disorders) | 0 | 3
Chills (General disorders) | 1 | 2
Energy increased (General disorders) | 2 | 3
Fatigue (General disorders) | 7 | 5
Irritability (General disorders) | 17 | 17
Thirst (General disorders) | 1 | 3
Hypersensitivity (Immune system disorders) | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 2
Rash pustular (Infections and infestations) | 0 | 3
Tooth abscess (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 17
Urinary tract infection (Infections and infestations) | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 1 | 4
Joint injury (Injury, poisoning and procedural complications) | 0 | 2
Joint sprain (Injury, poisoning and procedural complications) | 1 | 2
Skin laceration (Injury, poisoning and procedural complications) | 4 | 1
Thermal burn (Injury, poisoning and procedural complications) | 2 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 2
Weight increased (Investigations) | 1 | 7
Anorexia (Metabolism and nutrition disorders) | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Increased appetite (Metabolism and nutrition disorders) | 4 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Amnesia (Nervous system disorders) | 2 | 1
Disturbance in attention (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 7 | 8
Dysgeusia (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 18 | 15
Memory impairment (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 3
Somnolence (Nervous system disorders) | 11 | 8
Tremor (Nervous system disorders) | 3 | 4
Abnormal dreams (Psychiatric disorders) | 5 | 3
Agitation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 6 | 7
Depressed mood (Psychiatric disorders) | 5 | 4
Insomnia (Psychiatric disorders) | 17 | 10
Nightmare (Psychiatric disorders) | 3 | 3
Restlessness (Psychiatric disorders) | 3 | 2
Dysuria (Renal and urinary disorders) | 0 | 2
Pollakiuria (Renal and urinary disorders) | 3 | 2
Urine odour abnormal (Renal and urinary disorders) | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 6
Menstruation irregular (Reproductive system and breast disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acne (Skin and subcutaneous tissue disorders) | 4 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Hot flush (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.